CLINICAL TRIAL: NCT06197568
Title: An Open-Label, Safety, Tolerability and Efficacy Study of Vaginal AZU-101 in Postmenopausal Women
Brief Title: Open-Label Study of Vaginal AZU-101 in Postmenopausal Women
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Azure Biotech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GSM-201
Record Dates: First submitted 2023-12-05; First posted 2024-01-09 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Postmenopausal Symptoms
Keywords: Dyspareunia; Vaginal atrophy
MeSH Terms: conditions — Dyspareunia

STUDY DESIGN:
Intervention Model Description: Subjects will be enrolled into five cohorts (n=7/cohort).
Masking Description: This study is open-label. Randomization and blinding procedures will not be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Weekly 0.1 μg AZU-101 (Experimental): Weekly 0.1 μg vaginal dose of AZU-101
  Interventions: Drug: Lasofoxifene Tartrate (AZU-101)
- Weekly 0.5 μg AZU-101 (Experimental): Weekly 0.5 μg vaginal dose of AZU-101
  Interventions: Drug: Lasofoxifene Tartrate (AZU-101)
- Weekly 1 μg AZU-101 (Experimental): Weekly 1 μg vaginal dose of AZU-101
  Interventions: Drug: Lasofoxifene Tartrate (AZU-101)
- Twice-weekly 0.1 μg AZU-101 (Experimental): Twice-weekly 0.1 μg vaginal dose of AZU-101
  Interventions: Drug: Lasofoxifene Tartrate (AZU-101)
- Twice-weekly 0.5 μg AZU-101 (Experimental): Twice-weekly 0.5 μg vaginal dose of AZU-101
  Interventions: Drug: Lasofoxifene Tartrate (AZU-101)

INTERVENTIONS:
Drug: Lasofoxifene Tartrate (AZU-101) — 0.1 μg vaginal dose of AZU-101 weekly for 4 doses
  Other Names: AZU-101
  Arms: Weekly 0.1 μg AZU-101
Drug: Lasofoxifene Tartrate (AZU-101) — 0.5 μg vaginal dose of AZU-101 weekly for 4 doses
  Other Names: AZU-101
  Arms: Weekly 0.5 μg AZU-101
Drug: Lasofoxifene Tartrate (AZU-101) — 1 μg vaginal dose of AZU-101 weekly for 4 doses
  Other Names: AZU-101
  Arms: Weekly 1 μg AZU-101
Drug: Lasofoxifene Tartrate (AZU-101) — 0.1 μg vaginal dose of AZU-101 twice-weekly for 8 doses
  Other Names: AZU-101
  Arms: Twice-weekly 0.1 μg AZU-101
Drug: Lasofoxifene Tartrate (AZU-101) — 0.5 μg vaginal dose of AZU-101 twice-weekly for 8 doses
  Other Names: AZU-101
  Arms: Twice-weekly 0.5 μg AZU-101

SUMMARY:
Study Objectives:

Primary

° To evaluate the safety and tolerability of multiple vaginal doses of AZU-101 at 3 dose levels in postmenopausal women

Secondary

* To assess systemic pharmacokinetics (PK) of AZU-101
* To assess the efficacy of multiple vaginal doses of AZU-101 at 3 dose levels in postmenopausal women

DETAILED DESCRIPTION:
This is an open-label Phase 1b/2a study to evaluate the safety, pharmacokinetics (PK), and efficacy of vaginal AZU-101 in healthy postmenopausal female subjects over a period of 28 days. AZU-101 is a vaginal formulation of lasofoxifene tartrate, a selective estrogen receptor modulator (SERM).

A total of 35 subjects, age 45 to 65 years, will be assigned to five cohorts (Cohorts 1-5) sequentially during enrollment (n=7/cohort). A once-weekly dose of AZU-101 will be administered at a dose of 0.1 μg (Cohort 1), 0.5 μg (Cohort 2), or 1 μg (Cohort 3) for 4 doses. A twice-weekly dose of AZU-101 will be administered at a dose of 0.1 μg (Cohort 4) or 0.5 μg (Cohort 5) for 8 doses.

Safety and tolerability will be measured by vital signs, electrocardiogram (ECG) parameters, and the incidence of Treatment-Emergent Adverse Events (TEAEs) and concomitant treatments. The PK profile will be assessed using peak plasma concentration (Cmax), time to peak plasma concentration (tmax), and area-under-the-concentration-time-curve from time zero to infinity (AUC0-∞). Efficacy will be evaluated using vaginal pH, the vaginal Maturation Index (percentage of vaginal parabasal cells and superficial cells), and identification of the most bothersome symptom to the subject (dyspareunia, vaginal dryness, or vaginal irritation/itching).

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal female subjects between 45 and 65 years old, inclusive (at the time of signing informed consent) with at least:

   1. 12 months of spontaneous amenorrhea; or
   2. At least 6 weeks postsurgical bilateral oophorectomy.
2. Have self-identified at least one moderate to severe vaginal symptom that is most bothersome to her:

   1. Pain associated with sexual activity (dyspareunia)
   2. Vaginal dryness
   3. Vaginal irritation/itching
3. Vaginal pH ≥5.
4. Vaginal smear with the percentage of superficial cells not exceeding 5%
5. In the opinion of the Investigator, the subject will comply with the protocol and has a high probability of completing the study.

Exclusion Criteria:

1. Any contraindication to SERMs
2. Use of any of the following:

   1. Oral estrogen-, progestin-, androgen-, or SERM-containing drug products within 3 months before Screening Visit
   2. Transdermal hormone products within 4 weeks before Screening Visit
   3. Vaginal hormone products (rings, creams, gels) within 4 weeks before Screening Visit
   4. Intrauterine progestins within 8 weeks before Screening Visit
   5. Progestin implants/injectables or estrogen pellets/injectables within 6 months before Screening Visit
   6. Any medication, herbal product or nutritional supplement known or suspected to interact with AZU-101 within 2 weeks prior to Screening Visit
3. Evidence of underlying disease during the Screening Visit (performed within 28 days of Day 1) or at admission on Day 1.
4. A history or active presence of clinically important medical disease that might confound the study or be detrimental to the subject, including but not limited to:

   1. Endometrial hyperplasia
   2. Undiagnosed vaginal bleeding
   3. History of a chronic liver or kidney dysfunction/disorder (e.g., hepatitis C or chronic renal failure)
   4. Thrombophlebitis, thrombosis, or thromboembolic disorders
   5. Cerebrovascular accident, stroke, or transient ischemic attack
   6. Myocardial infarction or ischemic heart disease
   7. Malignancy or treatment for malignancy, within the previous 5 years, with the exception of basal cell carcinoma of the skin or squamous cell carcinoma of the skin
   8. History of estrogen dependent neoplasia, breast cancer, melanoma, or any gynecologic cancer, at any time
   9. Endocrine disease (except for controlled hypothyroidism or controlled non-insulin dependent diabetes mellitus)
   10. Known breast cancer gene (BRCA) mutation associated with increased risk of neoplasia
5. TVUS of the endometrium at Screening with a double-wall thickness measurement greater than 4 mm
6. Abnormal endometrial biopsy in non-hysterectomized women
7. A body mass index (BMI) <18 and >38 kg/m2
8. History of known alcohol or drug abuse within 1 year of the Screening Visit
9. Positive urine drug or alcohol screen at Screening Visit
10. Use of 15 or more cigarettes per day or current use of any electronic cigarettes
11. Use of an investigational drug or biologic within 60 days before administration of the first dose of study drug
12. Any clinically important abnormalities on Screening physical examination, assessments, ECG, or laboratory tests, including but not limited to:

    1. Unresolved cervical cytologic smear report of atypical glandular cells of undetermined significance (AGUS) or atypical squamous cells of undetermined significance (ASCUS). Cervical cytologic smear report of low-grade squamous intraepithelial lesion (SIL) or greater, cervical intraepithelial neoplasia (CIN) grade 1 or greater, or any reported dysplasia; Subjects with ASCUS are eligible only if high risk human papilloma virus (HPV) result is negative or she has a history of vaccination against HPV.
    2. Unresolved findings suspicious for malignancy on the breast exam; incomplete mammogram result (Breast Imaging Reporting and Data System [BI-RADS] category 0) or unresolved findings suggestive of malignant changes or findings requiring short interval follow-up on the pre-study mammogram (subjects must have mammography result of BI-RADS category 1 or 2 to enroll). Mammogram performed within 9 months prior to Screening Visit with documentation available may be used to evaluate study eligibility. The site must obtain a copy of the official report for the subject's study file, and it must be verified that the mammogram itself is available if needed for additional assessment.
    3. Hematocrit <35% or >45%
    4. Serum creatinine >15% of the upper limit of normal (ULN) for the laboratory used.
    5. Serum alanine aminotransferase (ALT) or serum aspartate aminotransferase (AST) >1.5 times the ULN for the laboratory used
    6. Fasting total cholesterol greater than 300 mg/dL (7.77 mmol/L) or triglycerides greater than 300 mg/dL (3.39 mmol/L)
    7. Positive laboratory finding for Factor V Leiden mutation
    8. Fasting glucose >125 mg/dL
    9. Uncontrolled hypertension (subjects with sitting BP >139 mmHg systolic or >89 mmHg diastolic) and may not be using more than 2 antihypertensive medications for the treatment of hypertension
    10. Uncontrolled hypotension; subjects with sitting BP <95 mmHg systolic or <65 mmHg diastolic
    11. A clinically significant abnormal 12-lead ECG (e.g., showing previous myocardial infarction or other findings suggestive of ischemia)
    12. Positive human immunodeficiency virus (HIV), hepatitis B, or hepatitis C

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 35 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Had Any Serious Adverse Events or Any Treatment Emergent Adverse Events With Severity Greater Than "Moderate" as measured by CTCAE v4.0 | 28 days
  Number of participants who had any serious adverse events or any adverse events with severity greater than "moderate," as determined by the Principal Investigator, using the composite safety assessment including clinical laboratory testing (full blood count, biochemistry, coagulation, lipid panel, thyroid hormone, urinalysis), ECG, vital signs, physical examination, transvaginal ultrasound, endometrial biopsy, and self-reporting of adverse events that are determined to be clinically significant.

SECONDARY OUTCOMES:
Pharmacokinetics (Cmax) | 24 hours after day 1
  Peak plasma concentration in pg/mL
Pharmacokinetics (Tmax) | 24 hours after day 1
  Time to peak plasma concentration in hours
Pharmacokinetics (AUC0-∞) | 24 hours after day 1
  Area under the concentration versus time curve in pg*hr/mL
Pharmacokinetics (Cmax) | 24 hours after day 21
  Peak plasma concentration in pg/mL
Pharmacokinetics (Tmax) | 24 hours after day 21
  Time to peak plasma concentration in hours
Pharmacokinetics (AUC0-∞) | 24 hours after day 21
  Area under the concentration versus time curve in pg*hr/mL
Efficacy (Vaginal pH) | 28 days
  Vaginal pH
Efficacy (Maturation index) | 28 days
  Ratio of percentage of superficial cells to percentage of basal cells
Efficacy (symptoms) | 28 days
  Change from baseline of the most bothersome symptom, as reported by the subject (pain associated with sexual activity, vaginal dryness, or vaginal irritation/itching), graded as 0=none; 1=mild; 2=moderate; 3=severe; range 0 to 3. Efficacy outcome will be proportion of subjects who improve at least one grade